CLINICAL TRIAL: NCT05401097
Title: Randomized, Sequential, Open-Label Study to Evaluate the Efficacy of IDH Targeted/Non- Targeted Versus Non-targeted/IDH-targeted Approaches in the Treatment of Newly Diagnosed IDH Mutated AML Patients Not Candidates for Intensive Induction Therapy (I- DATA Study)
Brief Title: IDH Targeted/Non- Targeted vs Non-targeted/IDH-targeted Approaches in the Treatment of Newly Diagnosed IDH Mutated AML Patients Not Candidates for Intensive Induction Therapy (I- DATA Study)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Alice Mims (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Alice Mims, Principal Investigator, Ohio State University Comprehensive Cancer Center
Organization: Ohio State University Comprehensive Cancer Center (Other)
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: OSU-21330; NCI-2022-01324 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); R01CA262496 (NIH)
Record Dates: First submitted 2022-05-16; First posted 2022-06-02 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Azacitidine; Biopsy; enasidenib; ivosidenib; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A (IDHi+Aza followed by Ven+aza) (Experimental): For IDH1 mutated AML patients randomized to first-line therapy with IDHi+aza, patients will receive Ivosidenib 500mg po orally daily on Days 1-28 of each 28 day cycle. For IDH2 mutated AML patients randomized to first-line therapy with IDHi+aza, patients will receive Enasidenib 100mg po orally daily on Days 1-28 of each 28 day cycle. Azacitidine will be given to both groups intravenously or subcutaneously at 75mg/m2 daily on days 1-7 or 1-5/8-9 of each 28 day cycle. Subsequent cycles after CR/CRi/CRh/MLFS achievement may be adjusted in timing and dosing.
  Interventions: Drug: Azacitidine; Procedure: Biopsy; Drug: Enasidenib; Drug: Ivosidenib; Drug: Venetoclax
- Arm B (Ven+aza followed by IDHi+aza) (Experimental): For both IDH1 and IDH2 mutated AML patient randomized to first-line therapy with Ven+aza, patients will receive venetoclax dosing with the ramp-up and dosing per the FDA-label (based off of concurrent drug interactions). Azacitidine will be given intravenously at 75mg/m2 daily on days 1-7 of each 28-day cycle. Subsequent cycles after CR/CRi/CRh/MLFS achievement may be adjusted in timing and dosing.
  Interventions: Drug: Azacitidine; Procedure: Biopsy; Drug: Enasidenib; Drug: Ivosidenib; Drug: Venetoclax

INTERVENTIONS:
Drug: Azacitidine — Given IV or SC
  Other Names: 5 AZC; 5-AC; 5-Azacytidine; 5-AZC; Azacytidine; Azacytidine, 5-; Ladakamycin; Mylosar; Onureg; U-18496; Vidaza
Procedure: Biopsy — Undergo biopsy of the bone marrow
  Other Names: BIOPSY_TYPE; Bx
Drug: Enasidenib — Given PO
  Other Names: AG-221; CC-90007 Free Base
Drug: Ivosidenib — Given PO
  Other Names: AG-120; Tibsovo
Drug: Venetoclax — Given PO
  Other Names: ABT-0199; ABT-199; ABT199; GDC-0199; RG7601; Venclexta; Venclyxto

SUMMARY:
This phase II study compares the order of treatment with ivosidenib or enasidenib and azacitidine plus venetoclax in treating older patients with acute myeloid leukemia with genetic changes in the IDH1 or IDH2 genes (IDH mutated). Ivosidenib is in a class of medications called isocitrate dehydrogenase-1 (IDH1) inhibitors. It works by slowing or stopping the growth of cancer cells. Enasidenib is in a class of medications called an IDH2 inhibitor. It also works by slowing or stopping the growth of cancer cells. Venetoclax is in a class of medications called B-cell lymphoma-2 (BCL-2) inhibitors. It may stop the growth of cancer cells by blocking Bcl-2, a protein needed for cancer cell survival. Azacitidine is in a class of medications called demethylation agents. It works by helping the bone marrow to produce normal blood cells and by killing abnormal cells. This study may help researchers determine which treatment order is best for older patients with IDH mutated acute myeloid leukemia: 1) ivosidenib or enasidenib followed by azacitidine plus venetoclax; or 2) azacitidine plus venetoclax followed by ivosidenib or enasidenib.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To compare overall treatment failure at 24 months in newly diagnosed IDH1 or IDH2 mutated AML patients ≥18 years who are not candidates for intensive induction chemotherapy randomized to either sequential treatment with an IDH inhibitor in combination with azacitidine followed by venetoclax in combination with azacitidine (Arm A) or sequential treatment with venetoclax in combination with azacitidine followed by an IDH inhibitor in combination with azacitidine (Arm B).

SECONDARY OBJECTIVES:

I. To compare overall survival at 24 months between patients treated on the two sequential treatment arms.

II. To compare time to overall treatment failure and time-to-event overall survival between patients treated on the two sequential treatment arms.

III. To determine the degree of response and compare complete remission (CR) rates, CR/complete remission with hematologic improvement (CRh)/complete remission with incomplete blood count recovery (CRi) rates, and overall response rates (CR/CRh/CRi/morphologic leukemia free state [MLFS]) for first-line therapy and second-line therapy between patients treated on the two sequential treatment arms.

IV. To compare the duration of response (CR/CRh/CRi) to first-line therapy and second-line therapy between patients treated on the two sequential treatment arms.

V. To determine toxicity profiles for patients treated on the two sequential treatment arms, overall and by first-line treatment and by second-line treatment.

VI. To determine causes that would not allow patients that first line treatment fails to go on to second line treatment.

VII. To determine the number and proportion of patients who are able to go onto allogeneic transplantation in both treatment arms.

EXPLORATORY OBJECTIVES:

I. To assess the clonal, biochemical and differentiation changes in AML cells during IDH-inhibitor and venetoclax treatment using flow cytometry and serial next generation sequencing on bone marrow specimens before and during treatment to assess for potential resistance mutations or clonal evolution that may be predictors of relapse.

II. To examine molecular properties of AML cells associated with primary and secondary resistance to each treatment arm to determine if particular subtypes of AML may be more or less likely to respond to a certain treatment modality.

III. To perform minimal residual disease (MRD) monitoring via liquid biopsy via our custom-designed 30-gene mutation ArcherPlex panel to monitor clonal dynamics during both sequential treatment arms.

IV. To determine the feasibility of longitudinal sociodemographic and social determinants of health (SDOH) data collection for adults with AML on a clinical trial.

V. To determine the acceptability of longitudinal sociodemographic/SDOH data collection for adults with AML on a clinical trial.

VI. To describe changes in SDOH for adults with AML on a clinical trial. VII. To describe associations between SDOH measures and trial outcomes for adults with AML on a clinical trial.

OUTLINE: Patients are randomized into 1 of 2 arms.

ARM A: For IDH1 mutated AML patients randomized to first-line therapy with IDHi+aza, patients will receive Ivosidenib 500mg po orally daily on Days 1-28 of each 28 day cycle. For IDH2 mutated AML patients randomized to first-line therapy with IDHi+aza, patients will receive Enasidenib 100mg po orally daily on Days 1-28 of each 28 day cycle. Azacitidine will be given to both groups intravenously or subcutaneously at 75mg/m2 daily on days 1-7 or 1-5/8-9 of each 28 day cycle. Subsequent cycles after CR/CRi/CRh/MLFS achievement may be adjusted in timing and dosing.

ARM B: For both IDH1 and IDH2 mutated AML patient randomized to first-line therapy with Ven+aza, patients will receive venetoclax dosing with the ramp-up and dosing per the FDA-label (based off of concurrent drug interactions). Azacitidine will be given intravenously at 75mg/m2 daily on days 1-7 of each 28-day cycle. Subsequent cycles after CR/CRi/CRh/MLFS achievement may be adjusted in timing and dosing.

After completion of the study treatment, patients are followed up at 30 days and then every 3 months for 5 years from registration, until death, or withdrawal of consent from study assessments and all further follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patients with newly diagnosed IDH1 or IDH2 mutated AML
* Not a candidate for or refuses intensive induction therapy
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Creatinine clearance > 40 ml/min
* Aspartate aminotransferase (AST)/ alanine aminotransferase (ALT) < 5 x upper limit of normal
* Total bilirubin < 1.5 x upper limit of normal (except for patients with Gilbert's disease)
* At the time of Venetoclax initiation, white blood cells (WBC) needs to be < 25 × 103 microliter: Hydroxyurea can be used to achieve that level.
* For female patients of childbearing potential, willingness to abstain from heterosexual intercourse or use a protocol-recommended method of contraception from the screening visit throughout the study treatment period and for 30 days following the last dose of either study drug. A serum pregnancy test will be done at screening. A serum or urine pregnancy test will be done on Day 1 of each cycle for women of childbearing potential. If the urine pregnancy test is positive, a serum pregnancy test must be performed per institutional standards.

The following methods are acceptable methods of contraception for the purpose of this study:

* Highly Effective Contraception Methods that can achieve a failure rate of less than 1% per year when used consistently and correctly are considered as highly effective birth control methods (Clinical Trials Facilitation Group 2014):

  * Combined (estrogen and progestin containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal, transdermal).
  * Progestin-only hormonal contraception associated with inhibition of ovulation (oral, injectable, implantable).
  * Intrauterine device.
  * Intrauterine hormone-releasing system.
  * Bilateral tubal occlusion.
  * Vasectomized partner, provided that partner is the sole sexual partner of the female study participant and that the vasectomized partner has received medical assessment of the surgical success.
  * Sexual abstinence- only if defined as refraining from heterosexual intercourse during the entire period of risk associated with the study treatments. The reliability of sexual abstinence needs to be evaluated in relation to the duration of the clinical study and the preferred and usual lifestyle of the patient.
* Acceptable Birth Control Methods that are not Highly Effective Contraception Acceptable birth control methods that result in a failure rate of more than 1% per year:

  * Progestin-only oral hormonal contraception, where inhibition of ovulation is not the primary mode of action.
  * Male or female condom with or without spermicide.
  * Cap, diaphragm, or sponge with spermicide. A combination of male condom with either cap, diaphragm, or sponge with spermicide (double barrier methods) are also acceptable, but not highly effective, birth control methods.
* The following methods are NOT acceptable methods of contraception for the purpose of this study:

  * Periodic abstinence (calendar, symptothermal, postovulation methods).
  * Withdrawal (coitus interruptus).
  * Spermicides only.
  * Lactational amenorrhea method.
  * Combination of male and female condom
* For male patients of childbearing potential having intercourse with females of childbearing potential, the willingness to abstain from heterosexual intercourse or use a protocol recommended method of contraception from the start of study treatment throughout the study treatment period and for 90 days following the last dose of either study drug. Males must also refrain from sperm donation from the start of study treatment throughout the study treatment period and for 90 days following the last dose of either dose of study drug

  * Willingness to comply with scheduled visits, drug administration plan, imaging studies, laboratory tests, other study procedures and study restrictions

Exclusion Criteria:

* Patients with acute promyelocytic leukemia
* Known active central nervous system involvement of leukemia
* History of active non-myeloid malignancy except for the following: adequately treated local basal cell carcinoma or squamous cell carcinoma of the skin, cervical carcinoma in situ, superficial bladder cancer, asymptomatic prostate cancer without known metastatic disease. patients receiving tamoxifen/Aromatase Inhibitors for non-metastatic breast cancer, or any other cancer that has been in complete remission without treatment for >= 5 years prior to enrollment
* Evidence of ongoing uncontrolled systemic bacterial, fungal or viral infection at the time of start of study treatment
* Uncontrolled infection with hepatitis C, hepatitis B, or human immunodeficiency virus (HIV)
* Pregnancy or breast feeding
* Concurrent participation in an investigational drug trial with therapeutic intent defined as prior study therapy within 14 days prior to study treatment
* Inability to tolerate oral medications including symptomatic disease significantly affecting gastrointestinal function such as inflammatory bowel disease or resection of stomach or small bowel

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Estimated)
Dates: Start 2022-09-13 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Overall treatment failure | At 12 months from date of randomization
  Defined as: 1) second occurrence of any of disease progression, relapse, failure to achieve complete remission (CR)/complete remission with hematologic improvement (CRh)/complete remission with incomplete blood count recovery (CRi), or 2) death from any cause. Within each treatment sequence, overall treatment failure rate will be defined as the number of patients with events divided by the number of eligible patients randomized. Patients who go to transplant will be considered a treatment success for a particular treatment sequence. All randomized patients meeting the eligibility criteria will be evaluable for treatment failure status by intention to treat. Will be analyzed using a Cochran-Mantel-Haenszel test, testing for a difference in proportions and stratifying on isocitrate dehydrogenase (IDH) mutation status.

SECONDARY OUTCOMES:
Difference in treatment failure rates between the two arms | Up to 2 years
  Will use a two-sided Cochran-Mantel-Haenszel test, stratifying on IDH mutation status.
Overall survival (OS) | Up to 5 years
  Will be summarized using the Kaplan-Meier method and will be compared between arms using a stratified log-rank test (stratified on IDH mutation status).
Duration of response | Up to 5 years
  Will be summarized using the Kaplan-Meier method and will be compared between arms using a stratified log-rank test (stratified on IDH mutation status).

CONTACTS AND LOCATIONS:
Overall Officials: Alice S Mims, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu